CLINICAL TRIAL: NCT02143817
Title: The Effect of Whole-body Vibration Training Combined With L-cit Supplementation on Cardiovascular, Autonomic Function and Body Composition in Postmenopausal Women
Brief Title: Whole Body Vibration Combined With L-citrulline Supplementation on Cardiovascular Function and Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: NOW Foods (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC2012.9674
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Pre-hypertension; Hypertension
Keywords: whole body vibration training; L-citrulline; hypertension; obesity; arterial function; arterial stiffness; autonomic function; endothelial function
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): This arm involves not making any change to the subject's lifestyle at the moment of the start of the intervention and for 8 wk.
- Whole body vibration training plus L-citrulline (Experimental): Lower-body exercise training on a vibration platform combined with L-citrulline supplemetation (6 grams/day)
  Interventions: Dietary Supplement: L-citrulline supplementation; Other: Whole Body Vibration Training
- Whole body vibration training & placebo (Experimental): Lower-body exercise training on a vibration platform combined with placebo supplementation (6 grams/day)
  Interventions: Other: Whole Body Vibration Training
- L-citrulline supplementation (Experimental): (6g per day)containing L-citrulline
  Interventions: Dietary Supplement: L-citrulline supplementation

INTERVENTIONS:
Dietary Supplement: L-citrulline supplementation
  Other Names: 8 weeks of L-citrulline supplementation in two doses of 3g each per day (6g per day)
  Arms: L-citrulline supplementation; Whole body vibration training plus L-citrulline
Other: Whole Body Vibration Training — The Whole body vibration training intervention consists of lower-body exercise in a vibration platform 3 times per wk for 8 wk. The subjects will perform static and dynamic exercises for the legs on the vibration platform. Dynamic exercises will be performed with slow controlled movements starting from an upright position into a 60 degree knee flexion (squat) and maximal heel elevation (toestand). Static exercises will be performed without movement in the joint angles described previously. The training volume will increase progressively over the 12-week training period by increasing the intensity of vibration, duration of the exercise set (30-60 sec), number of sets per exercise, and total duration of the training session, and decreasing the duration of rest periods (30-60 sec).The intensity of vibration and amplitude will also be increased progressively (25-30 Hz of frequency and from low to high amplitude).
  Arms: Whole body vibration training & placebo; Whole body vibration training plus L-citrulline

SUMMARY:
Arterial dysfunction contributes to the development of cardiovascular disease (CVD), which is currently afflicting millions of individuals. The use of the amino acid L-citrulline has been suggested as a potential aid for the treatment of CVD by increasing endothelial production of Nitric Oxide (NO). Whole body vibration (WBV) is new and effective form of exercise that is feasible for clinical populations and has been proven to decrease blood pressure (BP) and arterial stiffness and increase muscle mass and strength. Therefore, the purpose of this study was to investigate if the combination of WBV training (WBVT) plus L-citrulline supplementation would induce positive additive effects and would be an effective means to ameliorate arterial stiffness, endothelial function, BP and muscle strength/mass in postmenopausal women.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of 8 weeks combination of WBVT plus L-citrulline supplementation on arterial stiffness, endothelial function, BP and muscle strength/mass in overweight/obese postmenopausal women.

The specific aims of the study are:

1. To investigate if the additive effect of 8 weeks of WBVT combined with L-citrulline supplementation are more efficacious than either treatment alone in ameliorating cardiovascular disease risk factors by assessing arterial stiffness (aortic, systemic, and leg), aortic BP and wave reflection, and autonomic function (heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and baroreflex sensitivity). Flow mediated dilation and circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NO metabolites [NOx], 6-keto PGFIa, insulin, and ghrelin) and vasoconstrictors (endothelin-1 [ET-1],8-iso PGF2a,vascular endothelium growth factor [VGEF]) will be assessed as secondary outcome variables.
2. To evaluate the extent to which 8 weeks of WBVT combined with L-citrulline improves body composition assessed by changes in fat mass and lean mass using dual-energy x-ray absorptiometry and waist circumference.
3. To determine the additive effect of 8 weeks of WBVT combined with L-citrulline supplementation on muscle strength. These will be evaluated using the eight-repetition maximum test for the leg press and chest press exercises

ELIGIBILITY:
Inclusion Criteria:

Female 50 to 70 years of age At least 1 year after menopause Body mass index of 27-39.9 Sedentary or low active (less than 2 hr per wk)

Exclusion Criteria:

Younger than 50 or older than 70 years of age Body mass index lower than 27, or 40 or higher Physically active or competitively active Smoker Use of hormone replacement therapy of less than 1 yr Use of calcium channel blocker or beta blockers Use dietary supplementations (e.g.,L-arginine,L-citrulline,antioxidants) Uncontrolled diabetes Any restriction that would significantly interfere with compliance with the L-citrulline supplementation

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 8 weeks
  Non-invasive measures of brachial and aortic blood pressure
Arterial Stiffness and pressure wave reflection | 8 weeks
  Using pulse wave velocity of the aorta, systemic, and legs and the augmentation index from radial tonometry
Endothelial and autonomic functions | 8 weeks
  By measuring circulating levels of adipocytokines (adiponectin and leptin) and endothelial-derived vasodilators (NOx, 6-keto PGFIa, insulin, and ghrelin)and vasoconstrictors (ET-1 and 8-iso PGF2a, VEGF).In addition, heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and spontaneous baroreflex sensitivity will be assessed from electrocardiogram and beat-by-beat digital blood pressure.

SECONDARY OUTCOMES:
Body Composition | 8 weeks
  By measuring fat mass and lean soft tissue mass from dual-energy x-ray absorptiometry and waist circumference
Muscle Strength | 8 weeks
  Using eight-repetition maximum (8-RM) test for the leg press and chest press exercises

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Wong, Principal Investigator — Florida State University
Locations (1):
- FSU College of Human Sciences, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Wong A, Chernykh O, Figueroa A. Chronic l-citrulline supplementation improves cardiac sympathovagal balance in obese postmenopausal women: A preliminary report. Auton Neurosci. 2016 Jul;198:50-3. doi: 10.1016/j.autneu.2016.06.005. Epub 2016 Jun 24. PMID 27356482